CLINICAL TRIAL: NCT03879291
Title: Assessment of Utility of accelerateIQ in the Care of Patients Participating in a Pulmonary Rehabilitation Program
Acronym: GASSP
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: Karen Larimer (Industry)
Collaborators: Sunovian (Unknown)
Responsible Party: Sponsor-Investigator, Karen Larimer, Director of Clinical Development, physIQ, Inc.
Organization: physIQ, Inc. (Industry)
Other Study IDs: CTP-010
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: COPD; Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Other: pinpointIQ — The study will utilize physIQ's multivariate analytical methods that detect vital sign relationship changes compared to a patient's individual baseline. Changes in vital signs relationships may be indicative of current or future important clinical events. These changes are indicated through the Multivariate Change Index (MCI), which is a scalar index between 0 and 1, where values close to 0 indicate no significant change from baseline and values close to 1 indicated greater changes from baseline

SUMMARY:
The proposed study seeks to assess the performance of continuous biosensor data and machine learning analytics in assessment of health patient status in a pulmonary rehabilitation program.

It is hypothesized that using continuous physiologic biosensor data and machine learning analytics to detect changes in physiology may play a role in managing patients in the pulmonary rehabilitation setting.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 40 years of age;
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD);
* Enrolled in the study site's 12-week pulmonary rehabilitation program;
* Capable of completing a 6-minute walk test;
* Willing and able to comply with scheduled protocol procedures and follow up;
* Signed and dated informed consent and HIPAA materials indicating that the patient has agreed to participate in this study and has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

* Patient has cognitive or physical limitations that, in the opinion of the investigator, limit the patient's ability to utilize the System as instructed;
* Patient is actively enrolled in another clinical investigation that, in the opinion of the investigator, interferes with or compromises either that patient's ability to participation in this study or the ability for the study to generate results;
* Patients who have implanted defibrillators or pacemakers;
* Patient is allergic to hydrocolloid adhesive;
* Patient does not speak English.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be patients diagnosed with COPD participating in a pulmonary rehabilitation program.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical Utility | 90 days
  Correlation of reported health events with the multivariate change index

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore University Health System, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No